CLINICAL TRIAL: NCT00388141
Title: Nursing and Nurturing Premature Infants. An Intervention Study Investigating Systematic Use of Newborn Individualized Developmental Care Assessment Program NIDCAP® Improves Development of Infants and the Mothers' Parental Competence
Brief Title: Nursing and Nurturing Premature Infants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005 0149; NIDCAP, HAAG
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Infant Growth; Mothers' Parental Competence
Keywords: Preterm Infant;; NIDCAP;; Neonatal Care,; Intervention Study;; Growth and Development;; Maternal Self-esteem.; Maternal Social support; NICU
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIDCAP (Experimental): In the intervention NIDCAP group the staff has been introduced and trained in the principles of the NIDCAP-care, where main core is to see, organize and conduct the care of the preterm infant on behalf of the childs actually resources and competences
  Interventions: Behavioral: NIDCAP

INTERVENTIONS:
Behavioral: NIDCAP — Systematic care, where the mother and the nurses organize the caring on behalf of the preterm infants' ressources and developmental capacity such as the infant avoid over stimulation and distress
  Other Names: Newborn Individualized Developmental Care Assessment Program; Induvidualized Neonatal Care

SUMMARY:
The purpose of this study is to determine whether systematic use of the Newborn Individualized Developmental Care Assessment Program (NIDCAP®) improves the neurologic development of children and the parental competence of mothers.

DETAILED DESCRIPTION:
Background: The unborn infant's brain is growing from the fifth month of fetal life which makes preterm babies sensitive to environmental influence. Therefore, to prevent developmental brain injury is an essential goal for neonatal nurses.

Purpose: The study investigates whether systematic use of Newborn Individualized Developmental Care Assessment Program (NIDCAP®) improves the neurological development of preterm babies and the parental competence of mothers.

Design: This study compares postnatal care of preterm babies in two neonatal units.

Participants: Preterm infants born before 32 weeks' gestational age and their mothers.

Instruments:

* Preterm babies' behaviour in intervention and control groups is observed every 7-12 days using scoring sheets.
* Questionnaires focusing on maternal self esteem when the baby is 4 weeks and again at 3 and 18 months and 5 years.

Expected outcomes:

* Infants: less time with treatment using CPAP and oxygen, growth, time of discharge and pattern of motor behaviour.
* Mothers: self reported experiences of self esteem.

Analysis: t-test Expected implications: In a health promotion perspective the systematic NIDCAP program hopefully will constitute a more competent mother, knowledgeable in child care and parental management. The intervention NIDCAP®-care infant group is expected to increase in growth compared to the control group, their motor system will be more mature, and there will be an earlier discharge, all factors contributing positively to health economy.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants
* The infants' biological mothers

Exclusion Criteria:

* Premature infants with chromosomal anomaly
* Mothers who cannot read and understand Danish

Ages: 7 Days to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2005-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The mothers' self reported experiences of self esteem and social support | 18 months

SECONDARY OUTCOMES:
Infant growth | 18 months
Time of discharge | 18 months
Days of needing oxygen and respiratory support | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth OC Hall, Dr. med. PhD, Study Chair — University of Aarhus; Tine B Henriksen, MD, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Faculty of Health Science, University of Aarhus, Aarhus, Jylland, Denmark